CLINICAL TRIAL: NCT07025421
Title: The Arise Study - Use of Vertical Positioning
Acronym: ARISE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Peter Morris, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300014712; UAB (Other: University of Alabama at Birmingham)
Record Dates: First submitted 2025-06-09; First posted 2025-06-17 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Bed Position
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Upright bed positioning
  Interventions: Other: Intervention Upright Bed positioning
- Standard of Care (No Intervention): Standard of Care Head of Bed Elevation

INTERVENTIONS:
Other: Intervention Upright Bed positioning — Patient in receipt of the upright bed positioning will receive daily upright bed positioning time each day of mechanical ventilation following the time required by institutional protocol for ARDS - associated prone positioning
  Arms: Intervention

SUMMARY:
The pilot study will randomize 40 ARDS patients who if proning were required would be randomized to upright bed positioning or to stand of care with bed in the head of bed elevation position

DETAILED DESCRIPTION:
Patients will be randomized to receive either daily upright bed positioning or to receive standard of care with head of bed elevated.

ELIGIBILITY:
Inclusion Criteria:

- Acute Respiratory Distress Syndrome

Exclusion Criteria:

* Cancer
* Active tracheostomy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Tidal Volume | within first 7 days of mechanical ventilation
  Mechanical Ventilator Tidal Volume

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
Review with the UAB IRB for each request
Supporting Information: CSR
Time Frame: 2028 - 2030
Access Criteria: All credible research organizations - please contact the UAB Pulmonary Division office